CLINICAL TRIAL: NCT01375777
Title: A Randomized, Placebo- and Ezetimibe-controlled, Dose-ranging Study to Evaluate Tolerability and Efficacy of AMG 145 on LDL-C in Hypercholesterolemic Subjects With a 10-year Framingham Risk Score of 10% or Less
Brief Title: Monoclonal Antibody Against PCSK9 to Reduce Elevated Low-density Lipoprotein Cholesterol (LDL-C) in Adults Currently Not Receiving Drug Therapy for Easing Lipid Levels
Acronym: MENDEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101154
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hyperlipidemia
Keywords: High cholesterol; Proprotein convertase subtilisin/kexin type 9 (PCSK9); Treatment for high cholesterol; Lowering cholesterol; Lowering high cholesterol; Hypercholesterolemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia; Hypercholesterolemia, Autosomal Dominant, 3 | interventions — evolocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Placebo Q2W (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) for 12 weeks.
  Interventions: Other: Placebo to Evolocumab
- Placebo Q4W (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks (Q4W) for 12 weeks.
  Interventions: Other: Placebo to Evolocumab
- Ezetimibe (Active Comparator): Participants received 10 mg ezetimibe orally once a day for 12 weeks.
  Interventions: Drug: Ezetimibe
- Evolocumab 70 mg Q2W (Experimental): Participants received 70 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 105 mg Q2W (Experimental): Participants received 105 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 140 mg Q2W (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 280 mg Q4W (Experimental): Participants received 280 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 350 mg Q4W (Experimental): Participants received 350 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 420 mg Q4W (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab 105 mg Q2W; Evolocumab 140 mg Q2W; Evolocumab 280 mg Q4W; Evolocumab 350 mg Q4W; Evolocumab 420 mg Q4W; Evolocumab 70 mg Q2W
Drug: Ezetimibe — Administered orally once a day
  Other Names: Zetia
  Arms: Ezetimibe
Other: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: Placebo Q2W; Placebo Q4W

SUMMARY:
The primary objective was to evaluate the effect of 12 weeks of subcutaneous evolocumab (AMG 145) every 2 weeks (Q2W) or every 4 weeks (Q4W), compared with placebo, on the percent change from baseline in LDL-C when used as monotherapy in adults with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 75 years of age
* Low density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL and < 190 mg/dL
* Framingham risk score of 10% or less
* Fasting triglycerides < 400 mg/dL

Exclusion Criteria:

* History of coronary heart disease
* New York Heart Association (NYHA) II - IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2012-03-02 (Actual); Study Completion 2012-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (54):
- United States (37):
  - Research Site, Birmingham, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Encinitas, California
  - Research Site, Inglewood, California
  - Research Site, San Diego, California
  - Research Site, Tustin, California
  - Research Site, DeLand, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Sanford, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Brooklyn Center, Minnesota
  - Research Site, Las Vegas, Nevada
  - Research Site, Endwell, New York
  - Research Site, New Windsor, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Arlington, Texas
  - Research Site, Boerne, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Maroubra, New South Wales
  - Research Site, Carina Heights, Queensland
- Belgium (8):
  - Research Site, AnthÃ©e
  - Research Site, Dour
  - Research Site, Gozée
  - Research Site, Gribomont
  - Research Site, Halen
  - Research Site, Ham
  - Research Site, Linkebeek
  - Research Site, Retie
- Canada (4):
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, Toronto, Ontario
  - Research Site, Granby, Quebec
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle

REFERENCES:
- [Background] Koren MJ, Scott R, Kim JB, Knusel B, Liu T, Lei L, Bolognese M, Wasserman SM. Efficacy, safety, and tolerability of a monoclonal antibody to proprotein convertase subtilisin/kexin type 9 as monotherapy in patients with hypercholesterolaemia (MENDEL): a randomised, double-blind, placebo-controlled, phase 2 study. Lancet. 2012 Dec 8;380(9858):1995-2006. doi: 10.1016/S0140-6736(12)61771-1. Epub 2012 Nov 6. PMID 23141812
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adults 18 - 75 years with fasting low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL and < 190 mg/dL, fasting triglycerides ≤ 400 mg/dL and a National Cholesterol Education Program Adult Treatment Panel III Framingham risk score of 10% or less. First patient enrolled 06 July 2011, last patient enrolled 25 November 2011.
Pre-assignment Details: Participants were randomized with equal allocation into 1 of 9 treatment groups. Randomization was stratified on the basis of screening LDL-C concentration (< 130 mg/dL [3.4 mmol/L] or ≥ 130 mg/dL).
Period: Overall Study
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Started | 46 | 45 | 46 | 45 | 46 | 45 | 46 | 46 | 46
Received Treatment | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45
Completed | 44 | 42 | 45 | 45 | 45 | 44 | 44 | 44 | 44
Not Completed | 2 | 3 | 1 | 0 | 1 | 1 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of investigational product).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W | Total
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (9.8) | 50.7 (12.6) | 50.0 (12.0) | 50.9 (12.9) | 48.3 (11.8) | 52.8 (11.6) | 49.3 (10.3) | 50.9 (13.1) | 50.1 (12.0) | 50.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 26 | 30 | 33 | 36 | 28 | 33 | 26 | 267
  Male | 20 | 15 | 19 | 15 | 13 | 9 | 17 | 12 | 19 | 139
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Asian | 2 | 1 | 1 | 3 | 3 | 2 | 1 | 2 | 2 | 17
  Black or African American | 8 | 7 | 9 | 7 | 5 | 4 | 8 | 6 | 10 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  White | 35 | 36 | 35 | 33 | 37 | 39 | 35 | 36 | 33 | 319
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 6 | 5 | 5 | 5 | 8 | 7 | 5 | 10 | 56
  ot Hispanic or Latino | 40 | 39 | 40 | 40 | 41 | 37 | 38 | 40 | 35 | 350
Stratification Factor: LDL-C level [Number; unit: participants]
  < 130 mg/dL | 15 | 14 | 15 | 14 | 15 | 14 | 15 | 15 | 14 | 131
  ≥ 130 mg/dL | 30 | 31 | 30 | 31 | 31 | 31 | 30 | 30 | 31 | 275
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 147.0 (21.0) | 142.3 (24.3) | 144.2 (25.8) | 143.1 (21.7) | 141.5 (22.3) | 139.8 (21.1) | 141.1 (21.8) | 136.6 (20.8) | 138.9 (21.9) | 141.6 (22.3)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 173.8 (30.5) | 169.1 (27.7) | 170.0 (32.0) | 169.0 (24.5) | 169.2 (24.3) | 163.8 (23.7) | 166.3 (27.8) | 161.1 (26.1) | 167.9 (29.6) | 167.8 (27.4)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 111.7 (17.1) | 110.4 (17.2) | 109.9 (17.7) | 108.7 (15.7) | 108.5 (15.2) | 107.2 (16.3) | 109.2 (15.7) | 105.8 (15.9) | 110.2 (18.4) | 109.1 (16.5)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 4.477 (1.293) | 4.793 (1.836) | 4.670 (1.258) | 4.335 (1.090) | 4.571 (1.269) | 4.181 (1.131) | 4.500 (1.154) | 4.335 (1.282) | 4.741 (1.656) | 4.512 (1.351)
Apolipoprotein B/Apolipoprotein A-1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.729 (0.180) | 0.785 (0.322) | 0.752 (0.176) | 0.705 (0.161) | 0.744 (0.168) | 0.709 (0.175) | 0.751 (0.161) | 0.706 (0.185) | 0.758 (0.191) | 0.738 (0.196)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing ultracentrifugation (UC) LDL-C at Week 12 was imputed using last observation carried forward (LOCF) and calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45
percent change | -3.71 (2.66) | 4.54 (2.64) | -14.26 (2.60) | -40.98 (2.64) | -43.87 (2.60) | -50.93 (2.66) | -39.02 (2.57) | -43.20 (2.57) | -47.98 (2.58)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -47.23, 95% CI 2-sided [-54.52 to -39.93], Standard Error of Mean 3.70 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -40.17, 95% CI [-47.38 to -32.95], Standard Error of Mean 3.66 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -32.27, 95% CI 2-sided [-44.53 to -30.02], Standard Error of Mean 3.68 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -52.53, 95% CI 2-sided [-59.67 to -45.38], Standard Error of Mean 3.62 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -47.74, 95% CI 2-sided [-54.89 to -40.60], Standard Error of Mean 3.62 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -43.57, 95% CI 2-sided [-50.71 to -36.42], Standard Error of Mean 3.62 — Placebo is the reference

2. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing ultracentrifugation (UC) LDL-C at Week 12 was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45
mg/dL | -3.4 (3.9) | 7.3 (3.7) | -19.2 (3.6) | -55.7 (3.7) | -66.0 (3.7) | -69.3 (3.6) | -53.5 (3.6) | -56.7 (3.6) | -65.0 (3.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -65.9, 95% CI 2-sided [-76.3 to -55.6], Standard Error of Mean 5.2 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -62.7, 95% CI [-73.2 to -52.2], Standard Error of Mean 5.3 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -52.3, 95% CI 2-sided [-62.7 to -41.9], Standard Error of Mean 5.3 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -72.3, 95% CI 2-sided [-82.2 to -62.4], Standard Error of Mean 5.0 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -63.9, 95% CI 2-sided [-73.9 to -54.0], Standard Error of Mean 5.0 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -60.8, 95% CI 2-sided [-70.7 to -50.9], Standard Error of Mean 5.0 — Placebo is the reference

3. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45
percent change | -2.89 (2.40) | -0.25 (2.30) | -15.53 (2.36) | -37.95 (2.38) | -39.68 (2.34) | -48.04 (2.40) | -37.94 (2.24) | -42.14 (2.24) | -47.36 (2.25)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -45.15, 95% CI 2-sided [-51.72 to -38.58], Standard Error of Mean 3.33 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -36.79, 95% CI [-43.29 to -30.29], Standard Error of Mean 3.29 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -35.06, 95% CI 2-sided [-41.59 to -28.52], Standard Error of Mean 3.31 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -47.11, 95% CI 2-sided [-53.33 to -40.89], Standard Error of Mean 3.15 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -41.89, 95% CI 2-sided [-48.11 to -35.67], Standard Error of Mean 3.15 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -37.70, 95% CI 2-sided [-43.92 to -31.47], Standard Error of Mean 3.15 — Placebo is the reference

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45
percent change | -0.33 (2.28) | 0.19 (2.28) | -11.17 (2.19) | -32.66 (2.26) | -36.20 (2.23) | -44.52 (2.28) | -33.04 (2.21) | -37.73 (2.21) | -42.29 (2.22)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -44.19, 95% CI 2-sided [-50.45 to -37.94], Standard Error of Mean 3.17 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -35.87, 95% CI [-42.06 to -29.69], Standard Error of Mean 3.13 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -32.33, 95% CI 2-sided [-38.55 to -26.11], Standard Error of Mean 3.15 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -42.48, 95% CI 2-sided [-48.63 to -36.32], Standard Error of Mean 3.12 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -37.92, 95% CI 2-sided [-44.07 to -31.76], Standard Error of Mean 3.12 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -33.22, 95% CI 2-sided [-39.38 to -27.07], Standard Error of Mean 3.12 — Placebo is the reference

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45
percent change | -1.21 (2.17) | -3.39 (2.11) | -16.65 (1.99) | -30.07 (2.15) | -33.13 (2.12) | -38.70 (2.17) | -32.07 (2.05) | -34.60 (2.05) | -39.97 (2.06)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -37.49, 95% CI 2-sided [-43.43 to -31.54], Standard Error of Mean 3.01 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -31.92, 95% CI [-37.79 to -26.04], Standard Error of Mean 2.98 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -28.86, 95% CI 2-sided [-34.77 to -22.95], Standard Error of Mean 2.99 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -36.58, 95% CI 2-sided [-42.29 to -30.88], Standard Error of Mean 2.89 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -31.21, 95% CI 2-sided [-36.92 to -25.51], Standard Error of Mean 2.89 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -28.69, 95% CI 2-sided [-34.39 to -22.98], Standard Error of Mean 2.89 — Placebo is the reference

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A-1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 46 | 45 | 45 | 45 | 45
percent change | 2.03 (2.40) | 0.14 (2.46) | -12.35 (2.33) | -32.80 (2.38) | -38.30 (2.35) | -48.13 (2.40) | -36.10 (2.39) | -40.43 (2.39) | -45.33 (2.40)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -50.16, 95% CI 2-sided [-56.75 to -43.58], Standard Error of Mean 3.34 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -40.33, 95% CI [-46.84 to -33.82], Standard Error of Mean 3.30 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -34.83, 95% CI 2-sided [-41.38 to -28.28], Standard Error of Mean 3.32 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -45.47, 95% CI 2-sided [-52.12 to -38.82], Standard Error of Mean 3.37 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -40.57, 95% CI 2-sided [-47.22 to -33.92], Standard Error of Mean 3.37 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and the stratification factor; LS Mean Treatment Difference = -36.25, 95% CI 2-sided [-42.90 to -29.60], Standard Error of Mean 3.37 — Placebo is the reference

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo Q2W | Placebo Q4W | Ezetimibe | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45 | 0/45 | 1/46 | 1/45 | 0/45 | 1/45 | 0/45
Other Adverse Events (participants affected / at risk) | 10/45 | 10/45 | 14/45 | 11/45 | 11/46 | 14/45 | 7/45 | 11/45 | 9/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=45) | Placebo Q4W (N=45) | Ezetimibe (N=45) | Evolocumab 70 mg Q2W (N=45) | Evolocumab 105 mg Q2W (N=46) | Evolocumab 140 mg Q2W (N=45) | Evolocumab 280 mg Q4W (N=45) | Evolocumab 350 mg Q4W (N=45) | Evolocumab 420 mg Q4W (N=45)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=45) | Placebo Q4W (N=45) | Ezetimibe (N=45) | Evolocumab 70 mg Q2W (N=45) | Evolocumab 105 mg Q2W (N=46) | Evolocumab 140 mg Q2W (N=45) | Evolocumab 280 mg Q4W (N=45) | Evolocumab 350 mg Q4W (N=45) | Evolocumab 420 mg Q4W (N=45)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 2 | 0 | 2 | 0 | 3 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 2 | 0 | 1 | 3 | 0 | 1 | 2
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 4 | 2 | 2 | 1 | 1 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 5 | 3 | 2 | 2 | 3 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 1 | 1 | 2 | 1 | 1 | 3
Headache (Nervous system disorders) | 3 | 1 | 1 | 3 | 2 | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3 | 1 | 2 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 3 | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.